CLINICAL TRIAL: NCT03693222
Title: Effect of Quadratus Lumborum Block on Postoperative Analgesic Requirements in Pediatric Patients: A Randomized Controlled Double Blinded Study
Brief Title: Quadratus Lumborum Block in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BakirkoySadiKonuk
Record Dates: First submitted 2018-08-07; First posted 2018-10-02 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Pain
Keywords: Quadratus lumborum block, abdominal trunk block
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol; Morphine

STUDY DESIGN:
Intervention Model Description: Patients included in the study were randomly divided into 2 groups. Cases were assessed as intravenous opioid with 1 mg/kg tramadol HCl (Group O, n=20) or ultrasonography-guided quadratus lumborum block (Group B, n=20).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator's study is a prospective, randomized, double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tramadol use (Experimental): Cases were assessed as intravenous opioid with 1 mg/kg tramadol hydrochloride
  Interventions: Drug: Tramadol Hydrochloride; Drug: Morphine Sulfate
- quadratus lumborum block (Experimental): Cases were assessed asquadratus lumborum block for postoperative analgesia
  Interventions: Drug: Tramadol Hydrochloride; Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Tramadol Hydrochloride — The Wong-Baker facial pain scale was used to assess pain (1: no pain, 10: worst possible pain). During monitoring patients with pain score ≥3 had intravenous 1 mg/kg tramadol hydrochloride administered, After 15 minutes following tramadol injection, cases with pain score continuing ≥3 were to be assessed as insufficient analgesia and had 0.1 mg/kg morphine hydrochloride planned for intravenous administration.
Drug: Morphine Sulfate — The Wong-Baker facial pain scale was used to assess pain (1: no pain, 10: worst possible pain). During monitoring patients with pain score ≥3 had intravenous 1 mg/kg tramadol hydrochloride administered, After 15 minutes following tramadol injection, cases with pain score continuing ≥3 were to be assessed as insufficient analgesia and had 0.1 mg/kg morphine hydrochloride planned for intravenous administration.

SUMMARY:
Quadratus lumborum block (QLB) is a newly-defined trunk block performed with local anesthetic injection by imaging the abdominal muscles with ultrasonography (US) guidance; thus, analgesia is expected to be ensured from the T7-L1 dermatomal segment level.

In the study, the aim was to compare the postoperative analgesic effect of quadratus lumborum block in pediatric patients undergoing lower abdominal surgery

DETAILED DESCRIPTION:
Patients included in the study were randomly divided into 2 groups. Cases were assessed as intravenous opioid with 1 mg/kg tramadol HCl (Group O, n=20) or ultrasonography-guided quadratus lumborum block (Group B, n=20).

Total analgesic amounts in 24 hours and first analgesic requirement times recorded.

ELIGIBILITY:
Inclusion Criteria:

* The study included 40 cases undergoing lower abdominal surgery aged from 3 to 16 years with ASA (American Society of Anesthesiologist) I-II level.

Exclusion Criteria:

* Cases with ASA III-IV health level and those with a history of allergy to local anesthetic medications were not included in the study.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
postoperative total analgesic amounts in 24 hours | how many times in 24 hours
  the number of analgesic requirements

SECONDARY OUTCOMES:
first analgesic requirement times | in 24 hours
  first analgesic requirement times (hours)

IPD SHARING:
Plan to Share IPD: No